CLINICAL TRIAL: NCT03103698
Title: The Interest of the ANI in the Monitoring of Peroperative Analgesia in Bariatric Surgery: a Randomized Single Blind Study.
Brief Title: The Interest of the ANI in the Monitoring of Peroperative Analgesia in Bariatric Surgery
Acronym: ANI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2015_843_0032
Record Dates: First submitted 2017-03-31; First posted 2017-04-06 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Surgery; Obese
Keywords: analgesia per-operative
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monitoring of perioperative analgesia by the ANI device (Other)
  Interventions: Device: To demonstrate the monitoring of perioperative analgesia
- conventional monitoring based on hemodynamic variations. (Other)
  Interventions: Other: Standard preoperative evaluation of analgesia

INTERVENTIONS:
Device: To demonstrate the monitoring of perioperative analgesia — To demonstrate that the monitoring of perioperative analgesia by the ANI device decreases intraoperative morphine consumption compared with conventional monitoring based on haemodynamic variations.
  Arms: Monitoring of perioperative analgesia by the ANI device
Other: Standard preoperative evaluation of analgesia — To demonstrate that the monitoring of perioperative analgesia by the ANI device decreases intraoperative morphine consumption compared with conventional monitoring based on haemodynamic variations.
  Arms: conventional monitoring based on hemodynamic variations.

SUMMARY:
The intraoperative assessment of analgesia remains problematic and no analgesia monitor is used in routine practice.

DETAILED DESCRIPTION:
The intraoperative assessment of analgesia remains problematic and no analgesia monitor is used in routine practice. Currently, this assessment is based on hemodynamic changes, although hypertension or tachycardia is neither sensitive nor specific. An overdose in opioids exposes to many side effects ranging from respiratory depression to phenomena of post-operative hyperalgesia. Conversely, an under-dosage in opioids is at the origin of a nociceptive stress whose neurovegetative and hormonal response can aggravate post-operative morbidity or promote the occurrence of implicit memorization.

Nociceptive influx can not be detected directly. However, its ascent to the somesthetic area of the cerebral cortex leads to physiological reactions that can be evaluated. In particular, there are numerous anatomical and functional interactions between the autonomic nervous system and the nociceptive tract in the brain stem. These interactions are mainly at the level of the gray periqueducal substance, the rostral ventro-lateral bulbous region, the solitary tract nucleus and the hypothalamus. The nociceptive influx thus leads to changes in the activity of the ANS. The study of changes in the ANS would therefore be a method of assessing the intensity of the nociceptive influx.

This objective method can be used in the non-communicating or unconscious patient to evaluate the pain and to adapt the analgesic treatment to the best.

Obese patients who receive surgical management often have comorbidities such as restrictive syndrome, or obstructive sleep apnea syndrome. They thus represent a target of choice in perioperative analgesic optimization in order to avoid respiratory complications that may be related to over or under assay of morphine such as atelectasis, alveolar hypoventilation.

It is hypothesized that this device is more effective for the intraoperative evaluation of analgesia than the usual method based on hemodynamic changes in intraoperatively anesthetized patients for bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Major Patient Age ≥ 18 years
* Adult patients candidate for planned surgery with BMI> 30.
* Affiliation to social security.
* Patients who were clearly informed and signed consent.

Exclusion Criteria:

* Patient with a heart rhythm disorder.
* Respiratory rate less than 9 cycles / min.
* Irregular spontaneous ventilation.
* Perioperative use of a drug acting on the sinus node (eg atropine, etc.)
* History of neuropathic pain.
* Patient under morphine until the day before surgery.
* Patients under guardianship or curatorship or deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-10-17 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
The amount of morphine used per operatively in the two groups | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France